CLINICAL TRIAL: NCT04519268
Title: The Degree of Adherence of Pre-anesthetic Tests at Kasr Alaini Hospital to the NICE-UK Guidelines, and Its Effect on Decision Making & Patient Outcome: Prospective Observational Study
Brief Title: Adherence Degree of Kasr-Alaini Hospital Pre-anesthetic Tests to the NICE-UK Guidelines
Status: Completed | Type: Observational
Sponsor: Nazmy Edward Seif (Other)
Responsible Party: Sponsor-Investigator, Nazmy Edward Seif, Clinical Professor, Cairo University
Organization: Cairo University (Other)
Other Study IDs: ADPAT-KAH-NICEUKG
Record Dates: First submitted 2020-08-17; First posted 2020-08-19 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Anesthesia; Surgery; Exanimation
Keywords: Pre-anesthetic tests; NICE-UK guidlines; Kasr Alaini hospital
MeSH Terms: conditions — Coma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elective Surgical Adult Patients: Adult patients scheduled for an elective general surgical operation.
  Interventions: Diagnostic Test: Adult patients scheduled for an elective general surgical operation.

INTERVENTIONS:
Diagnostic Test: Adult patients scheduled for an elective general surgical operation. — The anesthesiologist, who is in charge of preoperative assessment at each hospital unit, will assess patients who are scheduled for elective surgery; and will inform senior anesthesiologists (with a minimum 3 years of experience) & consultant anesthesiologists, about the patients' data.
  Patients data with all requested preoperative investigations & required preparations, peri-operative course and post-operative outcome will be collected.

SUMMARY:
Routine preoperative tests aim to identify asymptomatic diseases that can't be recognized by history and examination. Identification and management of these diseases is thought to help minimizing perioperative morbidity and mortality. A large number of routine screening tests increase the cost of perioperative care. Also unneeded tests may harm the patient due to overtreatment for borderline / false positive results. Therefore, the routine use of such examinations remains controversial.

The National Institute of Health and Clinical Excellence (NICE-UK) guidelines for preoperative examination are the assessment standard developed by NICE in collaboration with the National Collaboration Center for Acute Care in the UK; in order to reduce unnecessary tests by recommending which tests should be offered to people before minor and major operations.

The aim of this study is to assess the degree of adherence of the current preoperative tests at Kasr Alaini hospital to the NICE guidelines, to assess the effectiveness and usefulness of the current practice of various examinations ordered by anesthesiologists during the pre-anesthetic evaluation in patients who are intended for elective surgery in the hospital and to also evaluate the cause of delay & its effect to predict postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients scheduled for elective surgical operations.

Exclusion Criteria:

* Patients operated upon an emergency basis.
* Pregnant females.
* Patients scheduled for cardio-thoracic and neurosurgical procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients that will be scheduled for an elective surgical operation at Kasr Alaini hospital during the study period.
Sampling Method: Probability Sample
Enrollment: 185 (Actual)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-01 (Actual)

PRIMARY OUTCOMES:
Degree of Adherence to NICE-UK Guidelines | one week
  The degree of adherence of the current practices at Kasr Alaini hospital preoperative testing to the NICE-UK guidelines, determined as a "percentage".

CONTACTS AND LOCATIONS:
Overall Officials: Beshoy A Naguib, MBBCh, Principal Investigator — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Nazmy S Michael, MD, Study Director — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University; Manar M Elkholy, MD, Study Chair — Kasr Al-Ainy Hospital, Faculty of Medicine, Cairo University
Locations (1):
- Cairo University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided